CLINICAL TRIAL: NCT03282799
Title: Pharmacokinetic and Pharmacodynamic Evaluation of Etonogestrel Dose Escalation With Efavirenz-based Antiretroviral Therapy in HIV-infected Ugandan
Brief Title: Pharmacologic Strategies for the Etonogestrel Implant in HIV-Infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine Anne Chappell (Other)
Collaborators: Infectious Disease Institute, Kampala, Uganda (Other); University of Nebraska (Other)
Responsible Party: Sponsor-Investigator, Catherine Anne Chappell, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17080453
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS; Contraception
Keywords: etonogestrel; efavirenz; antiretroviral therapy; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etonogestrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dose Etonogestrel Implant (Active Comparator): Single 68 mg etonogestrel implant
  Interventions: Drug: etonogestrel implant
- Increased Dose Etonogestrel Implant (Experimental): Two 68 mg (136 mg total) etonogestrel implants
  Interventions: Drug: etonogestrel implant

INTERVENTIONS:
Drug: etonogestrel implant — The etonogestrel implant is an contraceptive implant that is placed into the upper arm.
  Other Names: Nexplanon; Implanon

SUMMARY:
This study will evaluate the frequency of ovulation and cervical mucus quality of HIV-infected Ugandan women on efavirenz-based antiretroviral therapy using either a single etonogestrel implant or two etonogestrel implants for at least one year.

DETAILED DESCRIPTION:
This study is being done to compare the rate of ovulation when women receive two subdermal implant contraception devices containing the hormone etonogestrel (instead of only one device) while taking the HIV drug efavirenz. The etonogestrel implant is a device that is inserted under the skin on the upper arm and releases a small amount of drug into the body every day over a long period of time to prevent pregnancy for 3 years. A total of 72 non-pregnant women in Uganda, who agree to use the copper intrauterine device throughout the study, will participate in this study. Half will be assigned by chance to use one implant and half will be assigned to use two implants at the entry visit. After the entry visit to place the implant, visits will be scheduled 1 week, 4 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 21 weeks, 22, weeks, 23 weeks, 24 weeks, 36 weeks, 45 weeks, 46 weeks, 47 weeks, and 48 weeks after the implant(s) were placed. The rate of ovulation (determined by weekly endogenous progesterone concentrations in the blood during months 3, 6, and 12) will be compared between women that receive two 68 mg etonogestrel implants compared to one 68 mg etonogestrel implant in combination with efavirenz-based antiretroviral therapy. Cervical mucus quality (from cervical mucus samples collected weekly at months 3, 6, and 12), the blood concentration of etonogestrel (from blood samples collected at day 3 and weeks 1, 4, 12, 24, 36, 48) and efavirenz (from blood samples collected at enrollment and weeks 4, 12, 24, 36, 48, and the number of adverse events deemed related to etonogestrel implant use through 48 weeks will also be compared between the one- and two-implant study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Women aged 18 years to 40 years.
4. Diagnosed with HIV infection.
5. Medically eligible for the etonogestrel subdermal implant as a contraceptive method.
6. Receiving efavirenz-based anti-retroviral therapy for a minimum of 3 months prior to screening.
7. Must agree to have concurrent highly effective non-hormonal contraception with a copper intrauterine device, if not previously medically sterilized.
8. Participants must report regular menses (bleeding for 4-8 days at 21- to 35-day intervals) for the preceding 2 months.
9. Participants must have a negative urine pregnancy test at entry and report no unprotected sex since the last menstrual period or in the last two weeks.

Exclusion Criteria:

1. HIV RNA > 50 copies/mL at screening visit.
2. Serum hemoglobin < 10.0 g/dL.
3. Elevations in serum levels of alanine transaminase above 5 times the upper limit of normal.
4. Elevations in serum creatinine above 2.5 times the upper limit of normal.
5. Use of drugs known to be contraindicated with etonogestrel or efavirenz within 30 days of study entry. Due to the dynamic nature of drug interactions related to antiretroviral therapy, the study team will review all concomitant medications at screening for drug interactions with efavirenz and the etonogestrel implant.
6. Currently pregnant or postpartum less than 30 days at study entry.
7. Breastfeeding women within 6 months of delivery.
8. Use of hormonal contraception in the preceding 3 months prior to entry
9. Participants determined to be ineligible for intrauterine device placement.
10. Patients with a history of hypersensitivity to etonogestrel implant, undiagnosed vaginal bleeding, diagnosed or suspected sex hormone dependent neoplasia, benign or malignant liver tumor, or thromboembolic disease.
11. Presence of any active clinically significant disease or life-threatening disease that, in the investigator's opinion, would compromise the subject's safety or outcome of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Chappell, MD MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chappell CA, Lamorde M, Nakalema S, Kyohairwe I, Byakika-Kibwika P, Meyn LA, Pham MM, Scarsi KK. A randomized trial of double vs single-dose etonogestrel implant to overcome the interaction with efavirenz-based antiretroviral therapy. Am J Obstet Gynecol. 2024 Aug;231(2):242.e1-242.e9. doi: 10.1016/j.ajog.2024.03.001. Epub 2024 Mar 7. PMID 38458408

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Started | 36 | 36
Completed | 34 | 36
Not Completed | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 36] | 30 [29 to 35] | 31 [29 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ganda | 22 | 19 | 41
  Nkore | 5 | 1 | 6
  Nyarwanda | 2 | 3 | 5
  Soga | 2 | 1 | 3
  Tooro | 0 | 3 | 3
  Kiga | 1 | 3 | 4
  Other | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Uganda | 36 | 36 | 72
Weight [Median (Inter-Quartile Range); unit: kg] | 60.2 [54.0 to 69.1] | 59.2 [51.0 to 70.5] | 60.0 [52.6 to 69.4]
CD4+ cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 648 [602 to 923] | 700 [536 to 875] | 669 [547 to 880]
Prior live births [Median (Inter-Quartile Range); unit: births] | 3 [2.25 to 4] | 3 [2 to 3.75] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants That Ovulate During Month 3
Description: Proportion of participants that experience at least one ovulation during month 3 of etonogestrel implant use. Serum progesterone concentrations are measured weekly during month 3 (weeks 9-12). Ovulation is defined as endogenous progesterone concentrations of >3 ng/mL.
Time Frame: 3 months
Population: One participant in the standard dose arm was withdrawn at week 1 of the study due to pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
Participants | 11 | 0
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p < .001, Fisher Exact

2. Primary Outcome: Proportion of Participants That Ovulate During Month 6
Description: Proportion of participants that experience at least one ovulation during month 6 of etonogestrel implant use. Serum progesterone concentrations are measured weekly during month 6 (weeks 21-24). Ovulation is defined as endogenous progesterone concentrations of >3 ng/mL.
Time Frame: 6 months
Population: One participant in the standard dose arm was withdrawn at week 1 of the study due to pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
Participants | 17 | 0
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p < .001, Fisher Exact

3. Primary Outcome: Proportion of Participants That Ovulate During Month 12
Description: Proportion of participants that experience at least one ovulation during month 12 of etonogestrel implant use. Serum progesterone concentrations are measured weekly during month 12 (weeks 45-48). Ovulation is defined as endogenous progesterone concentrations of >3 ng/mL.
Time Frame: 12 months
Population: One participant in the standard dose arm was withdrawn at week 1 of the study due to pregnancy, and one was withdrawn at week 45 due to a mental health condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
Participants | 19 | 2
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p < .001, Fisher Exact

4. Secondary Outcome: Proportion of Cervical Mucus Scores Greater Than 10
Description: The proportion of World Health Organization cervical mucus scores that are greater than 10 from weekly samples collected during months 3, 6 and 12 of etonogestrel implant use. A cervical mucus score greater than 10 indicates the mucus is favorable for sperm penetration or lack of contraceptive effect. The cervical mucus score ranges from 0 indicating least favorable for sperm penetration to 15 for most favorable for sperm penetration.
Time Frame: 12 months
Population: Evaluable cervical mucus samples collected from participants over 48 weeks of etonogestrel implant use. One participant in the standard dose arm was withdrawn at week 1 of the study due to pregnancy.
Measure: Count of Units; unit: Cervical mucus samples
Units Other Than Participants: Cervical mucus samples
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
Number analyzed (Cervical mucus samples) | 249 | 234
Cervical mucus samples
  Cervical mucus score greater than 10 | 1 | 1
  Cervical mucus score of 10 or less | 248 | 233
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p > .99, Fisher Exact

5. Secondary Outcome: Median Efavirenz Concentration at Enrollment
Description: Median efavirenz concentrations measured in plasma samples collected at enrollment, prior to insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: Day 0
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
µg/mL | 2.26 [1.15 to 4.63] | 2.30 [1.28 to 3.65]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .685, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Median Efavirenz Concentration at Week 4
Description: Median efavirenz concentrations measured in plasma samples collected 4 weeks after insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: 4 weeks
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 and 1 participant who missed the 4-week visit.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
µg/mL | 2.41 [1.47 to 4.26] | 2.23 [1.38 to 5.46]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .784, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Median Efavirenz Concentration at Week 12
Description: Median efavirenz concentrations measured in plasma samples collected 12 weeks after insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: 12 weeks
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week and 1 participant who missed the 12-week visit.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
µg/mL | 2.10 [1.22 to 3.99] | 1.88 [1.35 to 2.87]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .587, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Median Efavirenz Concentration at Week 24
Description: Median efavirenz concentrations measured in plasma samples collected 24 weeks after insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: 24 weeks
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
µg/mL | 2.26 [1.31 to 4.12] | 1.76 [1.18 to 3.47]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .394, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Median Efavirenz Concentration at Week 36
Description: Median efavirenz concentrations measured in plasma samples collected 36 weeks after insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: 36 weeks
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
µg/mL | 1.97 [1.18 to 5.27] | 1.87 [1.09 to 4.28]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .660, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Median Efavirenz Concentration at Week 48
Description: Median efavirenz concentrations measured in plasma samples collected 48 weeks after insertion of the etonogestrel implant(s). Plasma efavirenz concentrations were quantified using a high-performance liquid chromatography assay with ultraviolet detection.
Time Frame: 48 weeks
Population: Efavirenz concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week and 1 participant who missed the 48-week visit.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
µg/mL | 2.05 [1.36 to 3.66] | 1.72 [1.01 to 2.73]
Statistical Analysis 1: Comparison: Standard Dose Etonogestrel Implant vs Increased Dose Etonogestrel Implant; Test type: Other; p = .290, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Median Etonogestrel Concentration at Week 1
Description: Median etonogestrel concentrations measured in plasma samples collected 1 week after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 1 week
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
pg/mL | 182 [102 to 303] | 439 [327 to 618]

12. Secondary Outcome: Median Etonogestrel Concentration at Week 4
Description: Median etonogestrel concentrations measured in plasma samples collected 4 weeks after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 4 weeks
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week and 1 participant who missed the 4-week visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
pg/mL | 115 [79 to 178] | 282 [158 to 414]

13. Secondary Outcome: Median Etonogestrel Concentration at Week 12
Description: Median etonogestrel concentrations measured in plasma samples collected 12 weeks after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 12 weeks
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week and 1 participant who missed the 12-week visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
pg/mL | 83 [66 to 99] | 214 [124 to 271]

14. Secondary Outcome: Median Etonogestrel Concentration at Week 24
Description: Median etonogestrel concentrations measured in plasma samples collected 24 weeks after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 24 weeks
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
pg/mL | 69 [41 to 99] | 168 [91 to 224]

15. Secondary Outcome: Median Etonogestrel Concentration at Week 36
Description: Median etonogestrel concentrations measured in plasma samples collected 36 weeks after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 36 weeks
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 35 | 36
pg/mL | 54 [42 to 71] | 132 [75 to 157]

16. Secondary Outcome: Median Etonogestrel Concentration at Week 48
Description: Median etonogestrel concentrations measured in plasma samples collected 48 weeks after insertion of the etonogestrel implant(s). Plasma etonogestrel concentrations were quantified using liquid chromatography tandem mass spectrometry.
Time Frame: 48 weeks
Population: Etonogestrel concentration not evaluated for 1 participant who was discontinued due to pregnancy at 1 week and 1 participant who missed the 48-week visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
Number analyzed (Participants) | 34 | 36
pg/mL | 39 [25 to 64] | 95 [69 to 137]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Standard Dose Etonogestrel Implant | Increased Dose Etonogestrel Implant
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 35/36 | 35/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Etonogestrel Implant (N=36) | Increased Dose Etonogestrel Implant (N=36)
Amenorrhea (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 23 (40) | 30 (68)
Metrorrhagia (Reproductive system and breast disorders) | 14 (20) | 22 (33)
Dysmenorrhea (Reproductive system and breast disorders) | 8 (10) | 10 (12)
Weight Gain (General disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 16 (26) | 15 (23)
Breast Tenderness (Reproductive system and breast disorders) | 1 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Implant Site Reaction (Product Issues) | 15 (19) | 24 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT03282799/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03282799/ICF_001.pdf